CLINICAL TRIAL: NCT02743546
Title: A Phase 1b Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of the Combination of Duvortuxizumab With Ibrutinib in Subjects With B-Cell Malignancies
Brief Title: Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Duvortuxizumab (JNJ-64052781) Plus Ibrutinib in Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108158; 64052781NHL1001 (Other: Janssen Research & Development, LLC); 2016-000721-39 (EudraCT Number)
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell
Keywords: B-Cell, Malignancy; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphocytic, Chronic, B-Cell; JNJ-64052781; Ibrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Neoplasms; Bronchiolitis Obliterans Syndrome | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Optimization:Participant with Certain B-Cell Malignancies (Experimental): Participants with certain B-cell malignancies (diffuse large B-cell lymphoma [DLBCL], mantle cell lymphoma [MCL], or follicular lymphoma [FL]) will receive rising doses of intravenous infusions of duvortuxizumab either with or without a priming dose in combination with oral ibrutinib until disease progression, unacceptable toxicity, or other protocol-specified withdrawal criteria are met. Dose escalation will continue until the recommended phase 2 dose or maximum tolerated dose is reached.
  Interventions: Drug: Duvortuxizumab; Drug: Ibrutinib
- Dose Expansion: Participants with DLBCL (Experimental): Participants with DLBCL will receive intravenous infusions of duvortuxizumab either with or without a priming dose in combination with oral ibrutinib at the recommended phase 2 dose until disease progression, unacceptable toxicity, or other protocol-specified withdrawal criteria are met.
  Interventions: Drug: Duvortuxizumab; Drug: Ibrutinib
- Dose Expansion: Participants with FL (Experimental): Participants with FL will receive intravenous infusions of duvortuxizumab either with or without a priming dose in combination with oral ibrutinib at the recommended phase 2 dose until disease progression, unacceptable toxicity, or other protocol-specified withdrawal criteria are met.
  Interventions: Drug: Duvortuxizumab; Drug: Ibrutinib
- Dose Expansion: Participants with MCL (Experimental): Participants with MCL will receive intravenous infusions of duvortuxizumab either with or without a priming dose in combination with oral ibrutinib at the recommended phase 2 dose until disease progression, unacceptable toxicity, or other protocol-specified withdrawal criteria are met.
  Interventions: Drug: Duvortuxizumab; Drug: Ibrutinib
- Dose Expansion: Participants with CLL (Experimental): Participants with chronic lymphocytic leukemia (CLL) will receive intravenous infusions of duvortuxizumab either with or without a priming dose in combination with oral ibrutinib at the recommended phase 2 dose until disease progression, unacceptable toxicity, or other protocol-specified withdrawal criteria are met.
  Interventions: Drug: Duvortuxizumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Duvortuxizumab — Duvortuxizumab will be administered at starting dose of 15 nanogram per kilogram (ng/kg) as an intravenous (IV) infusion during Part 1 (Dose Optimization) and at RP2D level determined in Part 1 during Part 2 (Dose Expansion). Participants will receive duvortuxizumab either with or without a priming dose. Participants who receive a priming dose will have infusions on Days 1, 8, and 22 of an initial 35-day cycle and then on Days 1 and 15 of 28-day cycles thereafter. Participants who do not receive a priming dose will have infusions on Days 1 and 15 of 28-day cycles.
Drug: Ibrutinib — Ibrutinib will be administered at 560 milligram per day (mg/day) orally once daily during Part 1 (Dose Optimization) and at a dose of 420 mg/day (for participants with CLL) or 560 mg/day (for participants with DLBCL, FL, or MCL) during Part 2 (Dose Expansion). In Part 1, ibrutinib will be initiated on Day 1 of the initial treatment cycle. In Part 2, ibrutinib will be initiated on Day -7 prior to the initial treatment cycle.

SUMMARY:
The purpose of this study is to determine whether duvortuxizumab and ibrutinib can be combined safely and to establish the maximum tolerated dose (MTD) in Part 1 and the recommended Phase 2 dose (RP2D) and to further explore the safety of duvortuxizumab in combination with ibrutinib at the RP2D in participants with diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), mantle cell lymphoma (MCL), and chronic lymphocytic leukemia (CLL) in Part 2.

DETAILED DESCRIPTION:
This is an open-label (identity of study drug will be known to participant and study staff), multicenter (when more than one hospital or medical school team work on a medical research study), Phase 1b study. The purpose of this study is to see if duvortuxizumab in combination with ibrutinib is safe and useful for treating participants with B-cell malignancies. This study will be conducted in 2 parts: Part 1: Dose Optimization and Part 2: Dose Expansion. Part 1 will determine what dose of duvortuxizumab can be given safely with the standard dose of ibrutinib to participants with previously treated B-cell malignancies. Part 2 will look at how previously treated DLBCL, FL, MCL, and CLL participants respond to a safe dose of duvortuxizumab in combination with ibrutinib. Part 2 will also test whether the dose from Part 1 is an effective cancer therapy. The study consists of a Screening Phase, an ibrutinib Run-In Phase (Part 2 only), a combination (duvortuxizumab plus ibrutinib) Treatment Phase (Day 1, Cycle 1 and continues until the completion of the End-of-Treatment Visit), End-of-Treatment Visit (30 days (+7 days) after the last dose of study drug), and Post-treatment Follow-up Phase. The end of the study will be defined as 12 months after the last participant has received the first dose of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a B-cell malignancy (diffuse large B-cell lymphoma [DLBCL], follicular lymphoma [FL], mantle cell lymphoma [MCL], or chronic lymphocytic leukemia [CLL]) with tumor progression following at least one (MCL and CLL) or two (DLBCL and FL) prior standard therapies
* The participant has a radiographically measurable tumor that requires treatment according to the treating physician
* The participant is able to carry out daily life activities with significant difficulty
* The participant has adequate organ and blood cell counts
* Sexually active participants must use medically acceptable methods of contraception during the course of the study

Exclusion Criteria:

* The participant has a brain tumor or significant side effects, including severe neurological side effects, from a previous anti-cancer treatment
* Current severe, uncontrolled systemic disease including an ongoing, active infection or history of clinically significant heart problems
* History of autoimmune disease, allogeneic hematopoietic stem cell transplant, or organ transplant
* The participant has received any of the following: ibrutinib or other Bruton's tyrosine kinase (BTK) inhibitor at any time; an agent targeting CD19-positive cells or CD3-expressing T cells at any time; or warfarin, a vitamin K antagonist, or a blood transfusion (red blood cells and/or platelets) within 1 week of starting the study
* The participant is pregnant, breastfeeding, or planning to become pregnant or father a child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-20 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose Limiting Toxicity | Approximately 9 months
  Dose limiting toxicity is based on adverse events and includes unacceptable hematologic toxicity, unacceptable non-hematologic toxicity, and laboratory abnormalities of Grade 4 or higher.
Part 1 and Part 2: Number of Participants With Adverse Events | Approximately 2 years
  An adverse event (AE) is any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship.
Part 1 and Part 2: Number of Participants With Serious Adverse Events | Approximately 2 years
  A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital abnormality.
Part 1 and Part 2: Change in Clinical Laboratory Values From Baseline | Baseline and 2 years
  Standard clinical chemistry and hematology panels will be used to evaluate changes in laboratory parameters in blood samples collected pre- and post-treatment.

SECONDARY OUTCOMES:
Part 1 and Part 2: Area Under the Serum Concentration-Time Curve From Time [0 to t] (AUC[0-t]) of Duvortuxizumab | Approximately 2 years
  The AUC[0-t] is the area under the duvortuxizumab serum concentration-time curve from time [0 to t].
Part 1 and Part 2: Area Under the Serum Concentration-Time Curve From Time [0 to t] (AUC[0-t]) of Ibrutinib | Approximately 2 years
  The AUC[0-t] is the area under the ibrutinib serum concentration-time curve from time [0 to t].
Part 1 and 2: Maximum Serum Concentration (Cmax) of Duvortuxizumab | Approximately 2 years
  The Cmax is the maximum observed serum concentration of duvortuxizumab.
Part 1 and 2: Maximum Serum Concentration (Cmax) of Ibrutinib | Approximately 2 years
  The Cmax is the maximum observed serum concentration of ibrutinib.
Part 1 and 2: Half-Life (t1/2) of Duvortuxizumab | Approximately 2 years
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration.
Part 1 and 2: Half-Life (t1/2) of Ibrutinib | Approximately 2 years
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration.
Part 1 and 2: Total Systemic Clearance (CL) of Duvortuxizumab | Approximately 2 years
  The CL is a quantitative measure of the rate at which duvortuxizumab is removed from the body.
Part 1 and 2: Total Systemic Clearance (CL) of Ibrutinib | Approximately 2 years
  The CL is a quantitative measure of the rate at which ibrutinib is removed from the body.
Part 1 and 2: Volume of Distribution at Steady-State (Vss) of Duvortuxizumab | Approximately 2 years
  The Vss is defined as the theoretical volume in which the total amount of duvortuxizumab would be uniformly distributed to produce the desired serum concentration of duvortuxizumab at steady state.
Part 1 and 2: Volume of Distribution at Steady-State (Vss) of Ibrutinib | Approximately 2 years
  The Vss is defined as the theoretical volume in which the total amount of ibrutinib would be uniformly distributed to produce the desired serum concentration of Ibrutinib at steady state.
Part 1 and Part 2: Number of Participants with Anti-Duvortuxizumab Antibodies | Approximately 2 years
  Plasma levels of antibodies to duvortuxizumab will be assessed for evaluation of potential immunogenicity.
Part 1 and Part 2: Objective Tumor Response | Approximately 2 years
  Objective tumor response is represented by participants who achieve a complete response (CR) or partial response (PR) to study treatment per the criteria for response assessment of Non-Hodgkin's Lymphoma (participants with diffuse large B-cell lymphoma [DLBCL], follicular lymphoma [FL], and mantle cell lymphoma [MCL]) or the International Workshop on chronic lymphocytic leukemia Criteria (IWCLL) (participants with CLL)
Part 1 and Part 2: Number of Participants With Complete Response (CR) | Approximately 2 years
  The CR rate is frequency of participants who achieve a complete response to study treatment according to the Criteria for Response Assessment of Non-Hodgkin's Lymphoma (participants with DLBCL, FL, and MCL) or the IWCLL Criteria (for participants with CLL).
Part 1 and Part 2: Duration of Response | Approximately 2 years
  The Duration of Response is defined as the time from the first observed response (CR or partial response [PR]) to documented disease progression or death due to any cause.
Part 1 and Part 2: 1-year Progression Free Survival (PFS) | 1 year
  Progression free survival is defined as the time from first enrollment into the study to documented disease progression or death due to any cause.
Part 1 and Part 2: 1-year Overall Survival | 1 year
  One-year survival is defined as the percentage of participants surviving 1 year after entering into the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC